CLINICAL TRIAL: NCT06030921
Title: Effects of State Trait Anxiety on Thorax, Diaphragm and Related Fascia.
Status: Completed | Type: Observational
Sponsor: The Touro College and University System (Other)
Responsible Party: Principal Investigator, Mikhail Volokitin, MD, DO., Principal Investigator, Associate Professor, The Touro College and University System
Other Study IDs: 16059
Record Dates: First submitted 2023-08-23; First posted 2023-09-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Anxiety State; Fascia; Anomaly
Keywords: Anxiety State, Fascial Strain, Osteopathic Medicine
MeSH Terms: conditions — Anxiety Disorders; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Osteopathic Structural Exam, State - Trait Anxiety Questionnaire — During a single patient encounter they will fill out the State-Trait Anxiety Questionnaire , and undergo a Osteopathic Structural Exam

SUMMARY:
Previous studies have accepted a strong correlation between anxiety and dysregulation in respiratory rate. The investigators would like to explore this correlation from an osteopathic perspective. The investigators seek to assess the muscles, bones, ligaments, and fascia related to the respiratory system, mainly the thoracic diaphragm. The study does not focus on clinically diagnosed General Anxiety Disorder but rather State-Trait Anxiety among medical student participants. State Anxiety is the temporary anxiety one feels in certain situations, and Trait Anxiety is the stable tendency to become anxious.

The investigators aim to assess somatic dysfunctions in medical students' respiratory systems and correlate those findings with their respective scores on the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) survey. The investigators will assess the patient's somatic dysfunction using an osteopathic structural exam, and the STICSA will quantify the patient's level of statetrait anxiety. This inquiry will further explore osteopathic medicine's perspective on addressing the patient as a whole by correlating the close relationship between one's mental state and the resultant physical dysfunctions within different areas of the body. Establishing this correlation can pave the way for a new perspective on treating mental health disorders that is both cost-effective and potentially more efficacious than the traditional method, which has a high relapse rate. Exploring the connection between somatic dysfunctions and state-trait anxiety will benefit the patient's overall well-being and add a new level of care that osteopathic physicians can provide to others.

DETAILED DESCRIPTION:
A common pattern in nature is that dysfunctions manifest in more than one way and on more than one canvas. For example, climate change is predicted to manifest as rising sea levels, warmer sea temperatures, destruction of coral reefs, droughts, and crop failure. This same pattern is seen physiologically as well. Osteopathic physicians commonly see a pattern of somatic dysfunctions secondary to a visceral pathology. Some viscerosomatic pathologies have predictable manifestations, seen as Chapman points, small tender nodules within deep fascia. This present study follows a similar investigation but attempts to connect the visceral emotion of anxiety with somatic dysfunctions seen in fascia. A growing body of literature has connected emotions to the physical body and the mechanism involved in this interconnectedness. This present study will not focus on elucidating new mechanisms, rather it will focus on using osteopathic medicine as the tool to assess the physical manifestations of state-trait anxiety.

Individuals with mental disorders have increased adverse health behaviors, higher rates of chronic medical conditions, and increased mortality. Out of all of the mental disorders, anxiety has the highest prevalence. A substantial percentage of students within health science programs ie. nursing, medicine, and pharmacy, have reported elevated scores on self-reported anxiety questionnaires during their first year. A recent study by Hoying et al. 2020 reported that 30% of graduate students in health science programs had elevated scores on self-reported anxiety measures when entering their first year. This is pertinent to the present study as most of the participants will be recruited from Touro COM's first-year OMS-I class. Additionally, most studies have focused on the clinical form of anxiety, such as generalized anxiety disorder, but few have thoroughly addressed the subclinical forms of anxiety. The present study focuses on state and trait anxiety as defined by Spileberger. State anxiety is the proclivity of one to perceive a situation as threatening and transiently experience apprehension, tension, and dread. Trait anxiety is the stable inclination to experience state anxiety to varying external stimuli.

Despite extensive research focused on the treatment of clinical forms of anxiety, remission rates remain low, most notably less than 50% remission in patients with a generalized anxiety disorder (GAD). The standard of care involves both pharmacologic and psychological modalities, but nevertheless, the desired outcome of complete remission is not achieved. Therefore, there is a push in the scientific community to investigate anxiety through the lens of alternative and complementary medicines (CAM). While this study does not propose a novel treatment modality for state-trait anxiety, it does propose a new lens through which state-trait anxiety can be assessed and further examined. Using osteopathic manipulative medicine, the examiners uncover physical manifestations of anxiety that might have been overlooked when using standard-of-care modalities. This study will examine how anxiety manifests in one's bones, muscles, ligaments, and other objective measures.

This study will focus exclusively on the thoracic (respiratory) diaphragm and related fascia to fully examine osteopathic medicine as a tool for assessing state-trait anxiety. The investigators believe that maximal convergence between the mechanisms that govern fascia, anxiety, and their physical manifestations is located within the thoracic fascia and its relationship to the diaphragm. Previous studies have explored the relationship between one's breathing rate and their measures on anxiety questionnaires. It is widely accepted that anxiety affects one's breathing rate and quality. To examine the related fascia to the thoracic diaphragm, the study will include structures enveloped by Sibson's fascia and the endothoracic fascia. These structures include muscles such as the sternocleidomastoid, anterior/posterior/middle scalene, external intercostals, pectoralis minor, and the thoracic diaphragm itself. The related bones include ribs 1 -12, the sternum, the xiphoid process, the L1-L3 vertebral bodies, and the L1-L3 Intervertebral disk. The ligaments include the right and left crus. Additionally, it is pertinent to measure subjects' respiratory rate, Co2 retention, diaphragmatic excursion, and any somatic dysfunctions found in their thoracic inlet or related to Zinc's common compensatory patterns. Assessment with osteopathic manipulative medicine is a viable, cost-effective, and sustainable solution for assessing anxiety.

Using the osteopathic structural exam, this study aims to correlate subjective and objective findings of measures stated above with participants' responses on the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) questionnaire. The STICSA inventory was chosen due to its superior ability to divide anxiety's cognitive and somatic aspects and distinguish state and trait anxiety. STICSA is also superior to the widely used State-Trait Anxiety Inventory in distinguishing between state-trait anxiety and depression.

This study is fundamental in furthering science's understanding of the intricate nature governing the mind-body connection. It is undeniable that one's psychological state influences one's physical well-being. Currently, there is a movement toward uncovering and exploring the biochemical, hormonal, and physiological interplay between the mind and the body. This study puts into action these discoveries and attempts to build a foundational framework on which future treatment modalities can be based. By examining state-trait anxiety through an osteopathic structural exam, focused on the thoracic diaphragm and its related fascial connection, this study attempts to quantify and qualify how state-trait anxiety manifests in one's body. If there is a significant result from our findings, it will call for many studies to replicate the results and, subsequently, future studies that use this foundation to find new ways to treat state-trait anxiety and potentially extrapolate these findings to different mental health diseases. This study has the potential to pivot the modern approach to assessing and treating mental health diseases. In addition, assessment with osteopathic manipulative medicine is a viable, cost-effective, and sustainable solution for assessing anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Touro College of Osteopathic Medicine Students of Harlem, Middletown, and Montana campus.
* Students from OMS-I to OMS-IV.
* Participants aged 18 - 45.

Exclusion Criteria:

* Previous history of generalized anxiety, depression, mania or hypomania, as defined by the DSM-IV, or a history of a bipolar mood disorder, personality disorder, or psychotic disorder.
* Presence of a cognitive disorder or dementia within 6 months before the baseline visit.
* Investigator believed there was a significant risk of suicide.
* Currently pregnant, lactating, o intending to become pregnant before, during, or within 30 days after participating in the study.
* Changes in medication use or psychotherapy during study period
* Presence of any other significant organic disease or serious illness (eg, cardiac, endocrine, gastrointestinal, infectious, liver or renal insufficiency, metabolic disturbance, neoplastic, neurologic, pulmonary, or vascular).
* Presence of any history of respiratory disorders including but not limited to asthma, COPD, emphysema
* History of abdominal or thoracic trauma or surgery within the past 10 years.
* Medication: Sympathomimetics, respiratory depressants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Touro College of Osteopathic Medicine Students, male and female, aged from 18-45.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Numerical scores collected from the STICSA survey | Through study completion, an average of 1 year.
  Numerical scores collected from the STICSA survey

SECONDARY OUTCOMES:
Quantity and Quality of Somatic Dysfunctions as examined by Osteopathic Structural Exam | Through study completion, an average of 1 year.
  Quantity and Quality of Somatic Dysfunctions as examined by Osteopathic Structural Exam

CONTACTS AND LOCATIONS:
Locations (1):
- Touro College of Osteopathic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Church JA. Climate change. How fast are sea levels rising? Science. 2001 Oct 26;294(5543):802-3. doi: 10.1126/science.1065714. PMID 11679657
- [Background] Ateweberhan M, McClanahan TR. Relationship between historical sea-surface temperature variability and climate change-induced coral mortality in the western Indian Ocean. Mar Pollut Bull. 2010 Jul;60(7):964-70. doi: 10.1016/j.marpolbul.2010.03.033. Epub 2010 May 5. PMID 20447661
- [Background] Bath M, Owens J. Physiology, Viscerosomatic Reflexes. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559218/ PMID 32644644
- [Background] Lookadoo RE, Bell JE. Public Health Policy Actions to Address Health Issues Associated with Drought in a Changing Climate. J Law Med Ethics. 2020 Dec;48(4):653-663. doi: 10.1177/1073110520979372. PMID 33404338
- [Background] Walker ER, McGee RE, Druss BG. Mortality in mental disorders and global disease burden implications: a systematic review and meta-analysis. JAMA Psychiatry. 2015 Apr;72(4):334-41. doi: 10.1001/jamapsychiatry.2014.2502. PMID 25671328
- [Background] Hoying J, Melnyk BM, Hutson E, Tan A. Prevalence and Correlates of Depression, Anxiety, Stress, Healthy Beliefs, and Lifestyle Behaviors in First-Year Graduate Health Sciences Students. Worldviews Evid Based Nurs. 2020 Feb;17(1):49-59. doi: 10.1111/wvn.12415. Epub 2020 Jan 8. PMID 31912989
- [Background] Mazurek Melnyk B, Slevin C, Militello L, Hoying J, Teall A, McGovern C. Physical health, lifestyle beliefs and behaviors, and mental health of entering graduate health professional students: Evidence to support screening and early intervention. J Am Assoc Nurse Pract. 2016 Apr;28(4):204-11. doi: 10.1002/2327-6924.12350. Epub 2016 Mar 16. PMID 26990269
- [Background] Endler NS, Kocovski NL. State and trait anxiety revisited. J Anxiety Disord. 2001 May-Jun;15(3):231-45. doi: 10.1016/s0887-6185(01)00060-3. PMID 11442141
- [Background] Spielberger, C. D. (1985a). "Anxiety, cognition and aﬀect: a state-trait perspective," in Anxiety and the Anxiety Disorders, eds A. H. Tuma, and J. D. Maser (Hillsdale, NJ: Lawrence Erlbaum Associates, Inc), 171-182
- [Background] Dixon L, Fotinos K, Sherifi E, Lokuge S, Fine A, Furtado M, Anand L, Liberatore K, Katzman MA. Effect of Osteopathic Manipulative Therapy on Generalized Anxiety Disorder. J Am Osteopath Assoc. 2020 Mar 1;120(3):133-143. doi: 10.7556/jaoa.2020.026. PMID 32091557
- [Background] Katzman MA, Bleau P, Blier P, Chokka P, Kjernisted K, Van Ameringen M; Canadian Anxiety Guidelines Initiative Group on behalf of the Anxiety Disorders Association of Canada/Association Canadienne des troubles anxieux and McGill University; Antony MM, Bouchard S, Brunet A, Flament M, Grigoriadis S, Mendlowitz S, O'Connor K, Rabheru K, Richter PM, Robichaud M, Walker JR. Canadian clinical practice guidelines for the management of anxiety, posttraumatic stress and obsessive-compulsive disorders. BMC Psychiatry. 2014;14 Suppl 1(Suppl 1):S1. doi: 10.1186/1471-244X-14-S1-S1. Epub 2014 Jul 2. PMID 25081580
- [Background] Ravindran AV, da Silva TL. Complementary and alternative therapies as add-on to pharmacotherapy for mood and anxiety disorders: a systematic review. J Affect Disord. 2013 Sep 25;150(3):707-19. doi: 10.1016/j.jad.2013.05.042. Epub 2013 Jun 12. PMID 23769610
- [Background] Ritz T, Meuret AE, Bhaskara L, Petersen S. Respiratory muscle tension as symptom generator in individuals with high anxiety sensitivity. Psychosom Med. 2013 Feb;75(2):187-95. doi: 10.1097/PSY.0b013e31827d1072. Epub 2013 Jan 16. PMID 23324873
- [Background] Wan HY, Stickford JL, Kitano K, Manz WJ, Koceja DM, Chapman RF, Stager JM. Acute hypercapnia does not alter voluntary drive to the diaphragm in healthy humans. Respir Physiol Neurobiol. 2018 Dec;258:60-68. doi: 10.1016/j.resp.2018.05.012. Epub 2018 May 30. PMID 29859322
- [Background] Bailey JE, Argyropoulos SV, Kendrick AH, Nash J, Jightman S, Nutt DJ. Inhalation of 35% CO2 results in subjective fear and activates the HPA axis in healthy volunteers. J Psychopharmacol. 2001;15:A22.
- [Background] Freire RC, Nardi AE. Panic disorder and the respiratory system: clinical subtype and challenge tests. Braz J Psychiatry. 2012 Jun;34 Suppl 1:S32-41. doi: 10.1590/s1516-44462012000500004. English, Portuguese. PMID 22729448
- [Background] Gilbert, C. (1998). Hyperventilation and the body. Journal of Bodywork and Movement Therapies, 2(3), 184-191
- [Background] Tindall IK, Curtis GJ, Locke V. Dimensionality and Measurement Invariance of the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) and Validity Comparison With Measures of Negative Emotionality. Front Psychol. 2021 Jun 7;12:644889. doi: 10.3389/fpsyg.2021.644889. eCollection 2021. PMID 34163400